CLINICAL TRIAL: NCT02432417
Title: A Phase II Randomized Controlled Trial for the Addition of Chloroquine, an Autophagy Inhibitor, to Concurrent Chemoradiation for Newly Diagnosed Glioblastoma
Brief Title: The Addition of Chloroquine to Chemoradiation for Glioblastoma,
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn due to a lack of funding. The researchers were unable to secure the necessary financial support to continue and complete the trial.
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLOROBRAINII
Record Dates: First submitted 2015-04-09; First posted 2015-05-04 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma; Astrocytoma, Grade IV
Keywords: Glioblastoma; Autophagy; EGFR; EGFRvIII; Chloroquine; Radiotherapy; Temozolomide
MeSH Terms: conditions — Glioblastoma | interventions — Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention): Radiotherapy and chemotherapy according to standard protocol for newly diagnosed GBM. This consists of 30 daily fractions of 2 Gray (Gy) or 33 daily fractions of 1.8 Gy to the tumor and surrounding margin in combination with TMZ 75 mg/m² Per os daily (po qd) and six adjuvant cycles of TMZ 150 - 200 mg/m² po qd.
- Experimental arm (Experimental): Radiotherapy and chemotherapy according to standard protocol for newly diagnosed GBM. This consists of 30 daily fractions of 2 Gray (Gy) or 33 daily fractions of 1.8 Gy to the tumor and surrounding margin in combination with TMZ 75 mg/m² Per os daily (po qd) and six adjuvant cycles of TMZ 150 - 200 mg/m² po qd.
  In addition this treatment will be combined with a daily intake of the recommended phase two dose (RPTD) of chloroquine (CQ).
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Chloroquine — CQ will start with one week before the start of radiotherapy and end on the last day of radiotherapy.
  Other Names: A-CQ
  Arms: Experimental arm

SUMMARY:
Glioblastomas (GBM) are the most common type of primary brain tumors with an annual incidence of approximately 500 patients in the Netherlands. Despite extensive treatment including a resection, radiation therapy and chemotherapy, the median overall survival is only 14.6 months.

Epidermal growth factor receptor (EGFR) amplification or mutation is regularly observed in GBM and is thought to be a major contributor to resistance to radiotherapy and chemotherapy. The most common EGFR mutation in GBM (EGFRvIII) is present in 30-50% of GBM.

Previously MAASTRO lab has shown that expression of EGFRvIII provides GBM cells with a survival advantage when exposed to stress factors such as hypoxia and nutrient deprivation. These metabolic stress factors activate a lysosomal degradation pathway, known as autophagy. Inhibition of autophagy sensitizes cells to hypoxia, reduces the viable hypoxic fraction in tumors with > 40% and subsequently sensitizes these tumors to irradiation.

Chloroquine (CQ) is a potent autophagy blocker and is the most widely investigated substance in this context. Previously, the effect of CQ has been demonstrated in a small randomized controlled trial in GBM treated with radiotherapy and carmustine. Although not statistically significantly different, the rate of death over time was approximately half as large in patients receiving CQ as in patients receiving placebo. The intracellular effects of CQ are dose-dependent. Therefore, the authors suggest an increase in daily dose of CQ may be necessary. Furthermore, the combination of CQ with TMZ may induce more damage to the neoplastic cells.

In the phase I part of this trial the recommended dose of CQ in combination with radiotherapy and temozolomide will be tested. In the phase II part of the trial patients with a histologically confirmed GBM will be randomized between standard treatment consisting of concurrent radiotherapy with temozolomide and adjuvant temozolomide (arm A) and standard treatment plus CQ (arm B).

DETAILED DESCRIPTION:
This study is a multi-centre randomized controlled, open label, phase II trial for patients with de-novo GBM.

Eligible patients will be randomized between arm A and arm B:

Arm A (standard): Radiotherapy and chemotherapy according to standard protocol for newly diagnosed GBM. This consists of 30 daily fractions of 2 Gy or 33 fractions in 1.8 Gy to the tumor and surrounding margin in combination with temozolomide 75 mg/m² per os daily (po qd) and six adjuvant cycles of temozolomide 150 - 200 mg/m² po qd.

Arm B (experimental): Standard treatment as described under arm A combined with daily intake of 400mg CQ. CQ will start with one week before the start of radiotherapy and end on the last day of radiotherapy.

In a single centre exploratory substudy, thirty subjects sequentially recruited within MAASTRO clinic randomized to arm B will be invited to receive two 3-[18F]fluoro- 2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1- yl)propan-1-ol PET-scans ([18F]HX4 ). The first on day -6 (start CQ), the second on day 0 (before the start radiotherapy and TMZ).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed grade IV supratentorial astrocytoma, IDH wildtype (glioblastoma multiforme)
* Tumor tissue available for histopathological analysis
* Diagnosis must have been made by biopsy or resection lower or equal than 3 months prior to study entry
* 18 - 70 years
* Karnofsky performance status greater or equal than 70
* Absolute neutrophil count at least 1.5 x 109/L and platelets at least 100 x109/L
* Adequate renal function
* Adequate hepatic function
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Females must have negative results for pregnancy tests performed
* No breast feeding.
* If male, subject must be surgically sterile or practicing a method of contraception
* Ability to swallow and take oral medication.

Exclusion Criteria:

* Prior radiotherapy
* Prior chemotherapy
* Pregnancy or breast feeding
* Recent (less than 3 months) severe cardiac disease (NYHA class greater than 1) (congestive heart failure, infarction)
* History of cardiac arrythmia (multifocal premature ventricular contractions, uncontrolled atrial fibrillation, bigeminy, trigeminy, ventricular tachycardia) which is symptomatic and requiring treatment, or asymptomatic sustained ventricular tachycardia. Asymptomatic atrial fibrillation controlled on medication is allowed.
* Cardiac conduction disturbances or medication potentially causing them
* Treatment with investigational drugs in 4 weeks prior to or during this study
* If the subject has clinically significant and uncontrolled major medical condition(s)
* Psychiatric illness/social situation that would limit compliance with study requirements
* Any medical condition, with the opinion of the study investigator, places the subject at an unacceptably high risk for toxicities.
* The subject has had another active malignancy within the past 3 years except for any cancer in situ that the principal Investigator considers to be cured.
* Chronic systemic immune therapy (with the exception of corticosteroids)
* Concurrent cytochrome P450 enzyme-inducing anticonvulsant drugs (e.g., phenytoin, carbamazepine, phenobarbital, primidone, or oxcarbazepine)
* Known glucose-6-phosphate dehydrogenase deficiency
* Psoriasis or porphyria
* Known hypersensitivity to 4-aminoquinoline compound
* Retinal or visual field changes unrelated to the tumor location prior to 4-aminoquinoline compound use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Six-month progression-free survival | Six months after start of study treatment
  The absence of documented disease progression (clinical or radiological) or death due to any cause within six months from randomization

SECONDARY OUTCOMES:
Overall survival | 2 years after start of study treatment
  Randomization until death by any cause
Adverse Events (AE) and serious AEs | 2 years after start of study treatment
  Acute and late toxic effects are scored according to Common Toxicity Criteria for Adverse Effects (CTCAE) 4.0
Gene mutation, deletion or amplification | 2 years
  O6-methylguanine-DNA-methyltransferase (MGMT), isocitrate dehydrogenase (IDH) and EGFRvIII in tumor tissue
Tumor hypoxia | Six months after start of study treatment
  Quantitative and qualitative assessment of [18F]HX4-PET obtained before treatment and one week after the start of CQ

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, prof., Principal Investigator — Maastro Clinic, The Netherlands

REFERENCES:
- [Background] Sotelo J, Briceno E, Lopez-Gonzalez MA. Adding chloroquine to conventional treatment for glioblastoma multiforme: a randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2006 Mar 7;144(5):337-43. doi: 10.7326/0003-4819-144-5-200603070-00008. PMID 16520474
- [Background] Jutten B, Keulers TG, Schaaf MB, Savelkouls K, Theys J, Span PN, Vooijs MA, Bussink J, Rouschop KM. EGFR overexpressing cells and tumors are dependent on autophagy for growth and survival. Radiother Oncol. 2013 Sep;108(3):479-83. doi: 10.1016/j.radonc.2013.06.033. Epub 2013 Jul 25. PMID 23891088
- [Background] Jutten B, Rouschop KM. EGFR signaling and autophagy dependence for growth, survival, and therapy resistance. Cell Cycle. 2014;13(1):42-51. doi: 10.4161/cc.27518. Epub 2013 Dec 13. PMID 24335351
- [Background] Rouschop KM, van den Beucken T, Dubois L, Niessen H, Bussink J, Savelkouls K, Keulers T, Mujcic H, Landuyt W, Voncken JW, Lambin P, van der Kogel AJ, Koritzinsky M, Wouters BG. The unfolded protein response protects human tumor cells during hypoxia through regulation of the autophagy genes MAP1LC3B and ATG5. J Clin Invest. 2010 Jan;120(1):127-41. doi: 10.1172/JCI40027. Epub 2009 Dec 14. PMID 20038797